CLINICAL TRIAL: NCT00542308
Title: An Open Label Single Arm Trial Investigating Zalutumumab, a Human Monoclonal Anti-EGF Receptor Antibody, in Combination With Best Supportive Care, in Patients With Non-Curable Squamous Cell Carcinoma of the Head and Neck Who Have Failed Standard Platinum-based Chemotherapy.
Brief Title: Zalutumumab in Non-curable Patients With SCCHN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GEN205
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Results first posted 2014-08-27 (Estimated); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Head and Neck Cancer; Squamous Cell Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms, Squamous Cell | interventions — zalutumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zalutumumab 4-16 mg/kg (Experimental): Zalutumumab iv infusion once weekly. The dose was titrated until grade 2 rash occurred.
  Interventions: Drug: Zalutumumab

INTERVENTIONS:
Drug: Zalutumumab — Individual dose titration weekly i.v. doses

SUMMARY:
Treatment, In combination with BSC, Open-label, Single arm, Efficacy Study.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age ≥ 18 years
2. Confirmed diagnosis, initially or at relapse, of squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx, considered incurable with standard therapy
3. Failure to at least one course of standard platinum-based chemotherapy

Exclusion Criteria:

1. Three or more prior chemotherapy regimens
2. Prior treatment with EGFr antibodies and/or EGFr small molecule inhibitors
3. Past or current malignancy other than SCCHN, except for certain other cancer diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steen Lisby, MD, Study Director — Genmab A/S, Bredgade 34, DK-1260 Copenhagen K, Denmark
Locations (48):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Loma Linda University Cancer Institute, Loma Linda, California
  - Moffitt Cancer Center, Tampa, Florida
  - Mountain States Tumor Institute, Boise, Idaho
  - University Of Chicago Medical Center, Chicago, Illinois
  - Ft. Wayne Medical Oncology/Hematology, Inc, Fort Wayne, Indiana
  - Henry Ford Health Systems, Detroit, Michigan
  - Oregon Health and Science University, Portland, Oregon
  - Baylor University Medical Center, Dallas, Texas
- Austria (3):
  - Medizinische Universität Graz, Graz
  - Universitätsklinik für Innere Medizin III, Salzburg
  - AKH Wien, Vienna
- Chile (3):
  - Instituto Clinico Oncologico del Sur ICOS, Temuco
  - Hospital Carlos Van Buren de Valparaiso, Valparaíso
  - Instituto Oncologico, Viña del Mar
- Colombia (4):
  - Centro de Investigaciones Oncologicas Clinica CIO San Diego S.A, Bogotá
  - Hospital Pablo Tobon Uribe, Medellín
  - Oncomedica S.A., Montería
  - Oncólogos del Occidente S.A., Pereira
- Czechia (4):
  - Facultni Nemocnice Hradec Kralove, Hradec Králové
  - Nemocnice Jihlava, Jihlava
  - Veseobecna Fakultni Nemocnice, Prague
  - Facultni Nemocnice Na Bulovce, Prague
- Germany (6):
  - Universitätsklinikum Essen, Essen
  - Klinikum der Johann Wolfgang Goethe Universität, Frankfurt am Main
  - Uniklinik Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Heidelberg, Heidelberg
  - Medizinische Universitätsklinik Lübeck, Lübeck
  - Südharz-Krankenhaus Nordhausen gGmbH, Nordhausen
- Israel (6):
  - Soroka Medical Center, Beersheba
  - Rambam Medial Center, Haifa
  - Shaare-Zedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
- Italy (3):
  - Istituto Nazionale Tumori, Milan
  - Istituto Europea di Oncologia, Milan
  - Azienda Ospedaliera Valtellina e Valchiavenna, Sondrio
- Peru (5):
  - Hospital Goyeneche, Arequipa
  - Hospital Nacional Carlos Alberto Seguin Escobedo, Arequipa
  - Hospital Nacional Almanzor Aguinaga Asenjo, Lambayeque
  - Hospital Central FAP, Lima
  - Hospital Nacional Guillermo Almenara Irigoyen, Lima
- Portugal (3):
  - IPO Coimbra, Coimbra
  - IPO Lisboa, Lisbon
  - IPO Porto, Porto
- Slovakia (2):
  - Narodny onkologicky ustav, Bratislava
  - FN Trnava, Trnava

REFERENCES:
- [Derived] Saloura V, Cohen EE, Licitra L, Billan S, Dinis J, Lisby S, Gauler TC. An open-label single-arm, phase II trial of zalutumumab, a human monoclonal anti-EGFR antibody, in patients with platinum-refractory squamous cell carcinoma of the head and neck. Cancer Chemother Pharmacol. 2014 Jun;73(6):1227-39. doi: 10.1007/s00280-014-2459-z. Epub 2014 Apr 9. PMID 24714973

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants attending Visit 2 were included in the FAS irrespective of their compliance with the planned course of zalutumumab.
Period: Overall Study
Arm/Group | Zalutumumab 4-16 mg/kg
Started | 90
Completed | 90
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants attending Visit 2 were included in the full analysis set irrespective of their compliance with the planned course of zalutumumab.
Arm/Group | Zalutumumab 4-16 mg/kg
Number analyzed (Participants) | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 70
  >=65 years | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 72
Region of Enrollment [Number; unit: participants]
  Portugal | 10
  United States | 22
  Czech Republic | 6
  Slovakia | 4
  Peru | 4
  Austria | 3
  Israel | 12
  Chile | 8
  Germany | 11
  Colombia | 1
  Italy | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as time from start of treatment until date of death of any cause.
Time Frame: From randomization until death, assessed up to 21 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Zalutumumab 4-16 mg/kg
Number analyzed (Participants) | 90
months | 5.3 [4.1 to 7.1]

2. Secondary Outcome: Objective Tumour Response
Description: Objective Tumour response according to Response Evaluation Criteria in Solid Tumours (RECIST v 1.0). Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the longest diameter of target lesions; Overall Response (OR), CR+PR. Stable disease is Responses not fulfilling CR, PR or progressive disease (PD). PD is At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started, OR the appearance of one or more new lesions.
Time Frame: During treatment and two weeks after end of treatment, assessed up to 21 months.
Population: All participants attending Visit 2 were included in the full analysis set irrespective of their compliance with the planned course of zalutumumab. Overall number of participants analyzed are number of participants with data available for analysis of best response.
Measure: Number; unit: participants
Arm/Group | Zalutumumab 4-16 mg/kg
Number analyzed (Participants) | 88
participants
  Complete response | 1
  Partial response | 4
  Stable response | 30
  Progressive disease | 33
  Not evaluable | 20

3. Secondary Outcome: Duration of Response
Description: DOR is defined among responders, as the time from the initial documentation of response to the date of disease progression or death, whichever occurs earlier.
Time Frame: During treatment and two weeks after end of treatment, assessed up to 21 months
Population: All participants attending Visit 2 were included in the full analysis set irrespective of their compliance with the planned course of zalutumumab. Overall number of participants analyzed are the number of participants with a response.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Zalutumumab 4-16 mg/kg
Number analyzed (Participants) | 5
days | NA [NA to NA] — Median and 95% confidence interval were not estimable due to insufficient number of participants with response.

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from start of treatment until disease progression or death.
Time Frame: During treatment and two weeks after end of treatment, assessed up to 21 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Zalutumumab 4-16 mg/kg
Number analyzed (Participants) | 90
months | 8.6 [8.0 to 10.4]

ADVERSE EVENTS:
Time Frame: From first dose until the end of the safety follow-up period (30 days after last dose) up to 93.58 weeks
Arm/Group | Zalutumumab 4-16 mg/kg
Serious Adverse Events (participants affected / at risk) | 83/90
Other Adverse Events (participants affected / at risk) | 90/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zalutumumab 4-16 mg/kg (N=90)
ANAEMIA (Blood and lymphatic system disorders) | 3 (3)
CARDIAC ARREST (Cardiac disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 5 (6)
OESOPHAGEAL FISTULA (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
DISEASE PROGRESSION (General disorders) | 55 (55)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 2 (3)
INFUSION RELATED REACTION (General disorders) | 1 (1)
OEDEMA (General disorders) | 1 (1)
PAIN (General disorders) | 1 (1)
PERFORMANCE STATUS DECREASED (General disorders) | 2 (2)
SUDDEN DEATH (General disorders) | 1 (1)
ABSCESS (Infections and infestations) | 1 (1)
CATHETER RELATED INFECTION (Infections and infestations) | 1 (1)
EYE INFECTION (Infections and infestations) | 1 (1)
LUNG INFECTION (Infections and infestations) | 2 (2)
PNEUMONIA (Infections and infestations) | 7 (8)
SEPSIS (Infections and infestations) | 1 (1)
SKIN INFECTION (Infections and infestations) | 1 (1)
SOFT TISSUE INFECTION (Infections and infestations) | 1 (1)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 (1)
UROSEPSIS (Infections and infestations) | 1 (1)
WOUND INFECTION (Infections and infestations) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (1)
WEIGHT DECREASED (Investigations) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 (4)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 4 (4)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1)
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 (1)
FACIAL PARESIS (Nervous system disorders) | 1 (1)
QUADRIPARESIS (Nervous system disorders) | 1 (1)
RENAL TUBULAR DISORDER (Renal and urinary disorders) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 9 (9)
HYDROPNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 3 (3)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2)
RESPIRATORY ACIDOSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zalutumumab 4-16 mg/kg (N=90)
ANAEMIA (Blood and lymphatic system disorders) | 10 (10)
CONJUNCTIVITIS (Eye disorders) | 6 (7)
CONSTIPATION (Gastrointestinal disorders) | 10 (10)
DIARRHOEA (Gastrointestinal disorders) | 12 (15)
NAUSEA (Gastrointestinal disorders) | 16 (22)
VOMITING (Gastrointestinal disorders) | 15 (20)
ASTHENIA (General disorders) | 17 (23)
FATIGUE (General disorders) | 19 (26)
MUCOSAL INFLAMMATION (General disorders) | 9 (12)
OEDEMA PERIPHERAL (General disorders) | 5 (5)
PAIN (General disorders) | 11 (14)
PYREXIA (General disorders) | 18 (31)
BRONCHITIS (Infections and infestations) | 7 (9)
FOLLICULITIS (Infections and infestations) | 6 (6)
PARONYCHIA (Infections and infestations) | 8 (8)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 (7)
HAEMOGLOBIN DECREASED (Investigations) | 8 (8)
WEIGHT DECREASED (Investigations) | 7 (8)
ANOREXIA (Metabolism and nutrition disorders) | 7 (8)
DECREASED APPETITE (Metabolism and nutrition disorders) | 6 (6)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 18 (26)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 7 (7)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 9 (10)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (8)
DIZZINESS (Nervous system disorders) | 5 (7)
HEADACHE (Nervous system disorders) | 16 (19)
INSOMNIA (Psychiatric disorders) | 10 (10)
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 (7)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 14 (16)
RHONCHI (Respiratory, thoracic and mediastinal disorders) | 5 (6)
PRURITUS (Skin and subcutaneous tissue disorders) | 10 (10)
RASH (Skin and subcutaneous tissue disorders) | 68 (85)
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 13 (14)
HYPERTENSION (Vascular disorders) | 5 (5)
HYPOTENSION (Vascular disorders) | 8 (8)

LIMITATIONS AND CAVEATS:
This was an uncontrolled single-arm open-label trial with no formal statistical tests planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The site and the PI may be required to withhold the publication for up to 90 days. Subject to a reasoned request from the sponsor, the publication may be further delayed for a period up to 6 months from the date of first submission to the sponsor.

The sponsor has the right to require deletion of any trade secret, proprietary, or confidential information supplied by the sponsor to the site or the PI. The sponsor shall not otherwise have the right to censor publications.